CLINICAL TRIAL: NCT06038149
Title: Improving Pulmonary Hypertension Screening by Echocardiography
Acronym: IMPULSE
Status: Recruiting | Type: Observational
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); Royal Free Hospital NHS Foundation Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Royal Papworth Hospital (Other Government); Golden Jubilee National Hospital (Other Government); University of Bath (Other); Liverpool John Moores University (Other)
Responsible Party: Sponsor
Other Study IDs: IMPULSE
Record Dates: First submitted 2023-06-21; First posted 2023-09-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low PH probability: Individuals identified as being of a low risk of pulmonary hypertension on routine echocardiography through existing British Society of Echocardiography/ European Society of Cardiology guidelines will undergo a research echocardiogram on the day of their planned right heart catheter.
  Interventions: Diagnostic Test: Transthoracic echocardiogram
- Intermediate PH probability: Individuals identified as being of an intermediate risk of pulmonary hypertension on routine echocardiography through existing British Society of Echocardiography/ European Society of Cardiology guidelines will undergo a research echocardiogram on the day of their planned right heart catheter.
  Interventions: Diagnostic Test: Transthoracic echocardiogram

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiogram — A painless ultrasound scan of the heart.
  Other Names: TTE

SUMMARY:
This study aims to assess the application of the novel IMPULSE algorithm for the detection of pulmonary hypertension (PH) in those with a low or intermediate probability of PH according to the British Society of Echocardiography (ESC) and European Society of Cardiology (ESC) guidelines.

DETAILED DESCRIPTION:
This is a prospective, multi-centre cross-sectional study with a planned 18 month longitudinal component.

Participants will be recruited from patients referred for the first time for transthoracic echocardiography at the Royal United Hospitals Bath National Health Service (NHS) Foundation Trust, Royal Free Hospital NHS Foundation Trust, Sheffield Teaching Hospitals, Royal Papworth Hospital, and Golden Jubilee Hospital.

The investigators will prospectively recruit patients without a diagnosis of Pulmonary Hypertension.

Transthoracic echocardiographic (TTE) imaging will be performed in line with British Society of Echocardiography minimum dataset guidelines, and comprehensive right heart echocardiographic imaging and analysis will be performed following the British Society of Echocardiography recommendations for assessing right heart function, in addition to the IMPULSE algorithm;

A right ventricular free wall longitudinal strain value of less than -23%, or, right ventricular fractional area change (FAC) less than 35% in females/30% in males, in addition to a right ventricular isovolumetric relaxation time in excess of 73ms in patients with low/Intermediate probability of PH by current guidelines would categorise that patient as being IMPULSE positive.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained breathlessness
* Risk factors for Pulmonary arterial hypertension (PAH), chronic thromboembolic pulmonary hypertension (CTEPH)
* Unexplained elevation of B-type natriuretic peptide (BNP/proBNP)
* Referred for catheterisation.

Exclusion Criteria:

* ESC / BSE echo high probability of PH
* Known or suspected congenital heart disease
* Patients unlikely to benefit from management of PH or its underlying causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred into a UK pulmonary hypertension centre for the first time, determined to be of low/intermediate probability of pulmonary hypertension on routine echocardiogram.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Analysis of the IMPULSE algorithm in the assessment of pulmonary hypertension | 18 months
  Analyse sensitivity, specificity, positive predictive value, negative predictive value, accuracy of IMPULSE algorithm on the assessment of PH.
Analysis of the IMPULSE algorithm in comparison to existing guidlines | 18 months
  Analyse sensitivity, specificity, positive predictive value, negative predictive value, accuracy of IMPULSE algorithm in comparison with the existing ESC PH guidelines.

SECONDARY OUTCOMES:
Analysis of additional echocardiographic measurements of right heart systolic function not utilised in the assessment of pulmonary hypertension. | 18 months
  Values from echocardiographic measures of right heart systolic function not currently used in the ESC/BSE echocardiography pulmonary hypertension, or IMPULSE algorithms will be analysed for sensitivity, specificity, positive predictive value and negative predictive value in context with with values obtained during formal pulmonary hypertension diagnosis via right heart catheter, in patients already found to have a mild to intermediate probability of pulmonary hypertension.
Analysis of additional echocardiographic measurements of right heart diastolic function not utilised in the assessment of pulmonary hypertension. | 18 months
  Values from echocardiographic measures of right heart diastolic function not currently used in the ESC/BSE echocardiography pulmonary hypertension, or IMPULSE algorithms will be analysed for sensitivity, specificity, positive predictive value and negative predictive value in context with with values obtained during formal pulmonary hypertension diagnosis via right heart catheter, in patients already found to have a mild to intermediate probability of pulmonary hypertension.
Analysis of additional echocardiographic measurements of left heart function not utilised in the assessment of pulmonary hypertension. | 18 months
  Values obtained in the echocardiographic assessment of left heart disease not currently used in the ESC/BSE echocardiography pulmonary hypertension, or IMPULSE algorithms will be analysed for sensitivity, specificity, positive predictive value and negative predictive value in context with values obtained during formal pulmonary hypertension diagnosis via right heart catheter, in patients already found to have a mild to intermediate probability of pulmonary hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel X Augustine, BSc(Hons), Principal Investigator — Royal United Hospitall NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Royal United Hospital NHS Foundation Trust, Bath, Banes
  - Golden Jubilee Hospital, Glasgow, Lanarkshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - Royal Papworth Hospital, Cambridge
  - Royal Free NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Study documentation will be disseminated to all participating sites on approval.
  All research echocardiography data will be transferred to the core lab in the Royal United Hospital Bath for analysis.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data obtained will be made available during the data collection period and transferred in batches.
Access Criteria: Transfer via internal NHS DICOM servers